CLINICAL TRIAL: NCT04255875
Title: A RANDOMIZED, DOUBLE-BLIND, PLACEBO CONTROLLED EVALUATION OF SINGLE DOSES OF PF-07209326 IN HEALTHY PARTICIPANTS (SAFETY, TOLERABILITY, AND PHARMACOKINETICS [PK]) FOLLOWED BY AN OPEN LABEL, REPEAT DOSE EVALUATION IN SICKLE CELL DISEASE PARTICIPANTS (SAFETY, TOLERABILITY, PK AND EFFICACY)
Brief Title: Dose Escalation Study of PF-07209326 in Healthy Participants and Participants With Sickle Cell Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: C4071001
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Healthy; Sickle Cell Anemia
Keywords: Safety; Tolerability; Single ascending dose; Multiple dose; Pharmacokinetics; Phase 1; First in human; First in patient
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Masking will only be applicable to Part 1 of the study where Healthy participants will be enrolled and randomized to receive either PF-07209326 or to placebo. In Part 2 of the study, all eligible SCD participants will receive PF-07209326 and no masking will be required.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment Healthy Participants (Experimental): Participants will receive single ascending doses of subcutaneous (SC) or intravenous PF-07209326
  Interventions: Biological: PF-07209326
- Placebo Healthy Participants (Placebo Comparator): Participants will receive matching placebo
  Interventions: Biological: Placebo
- Treatment for SCD (Experimental): Participants will receive a multiple dose of subcutaneous PF-07209326
  Interventions: Biological: PF-07209326

INTERVENTIONS:
Biological: Placebo — Participants will receive matching placebo
  Arms: Placebo Healthy Participants
Biological: PF-07209326 — Participants will receive SC or IV single ascending doses
  Arms: Treatment Healthy Participants
Biological: PF-07209326 — SCD participants will receive a multiple dose of subcutaneous PF-07209326
  Arms: Treatment for SCD

SUMMARY:
This Phase 1 first-in-human, first-in-patient, single ascending dose and multiple dose study will be a randomized, double-blind, placebo-controlled investigation of the safety, tolerability, and pharmacokinetics of PF-07209326 in healthy participants and participants with sickle cell disease.

DETAILED DESCRIPTION:
Part 1 will evaluate the safety and tolerability, pharmacokinetics and pharmacodynamics of single ascending doses of PF-07209326 delivered by subcutaneous injection or intravenous delivery in healthy volunteer participants. After establishing the safety and tolerability in healthy participants, Part 2 will evaluate the safety and tolerability, pharmacokinetics and pharmacodynamics of subcutaneously delivered multiple dose of PF-07209326 in participants with sickle cell disease.

ELIGIBILITY:
Inclusion Criteria Health Participants:

1. Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria Healthy Participants:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, immunocompromised (or known disorder of the immune system), cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C antibody (HCVAb). Hepatitis B vaccination is allowed.
3. History of active or latent tuberculosis (TB) regardless of treatment or positive QuantiFeron TB test.
4. Participants with any of the following acute or chronic infections or infection history:

   * Any infection requiring treatment within 2 weeks prior to the screening visit.
   * Any infection requiring hospitalization, parenteral antimicrobial therapy within 30 days of the first dose of investigational product.
   * Any infection judged to be an opportunistic infection, within the past 6 months of the first dose of the investigational product.
   * Known active or history of frequent bacterial, viral, fungal, mycobacterial or other infections as determined by the PI.
   * Participants with a fever within the last 7 days prior to dosing.
5. Participants with a history of allergic or anaphylactic reaction to therapeutic or diagnostic protein.
6. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.

Inclusion Criteria for SCD Participants

1. Participants between the ages of 16 and 70 years old with a confirmed diagnosis of stable sickle cell disease (HbSS or HBS β0 thalassemia).
2. Medical history of ≥2 and ≤ 10 medical utilization VOCs in 12 months prior to screening.
3. ≥75% of daily ePRO diary completion, over a minimum of 14 days during the screening period.
4. Fully vaccinated for COVID-19 in accordance with the Center for Disease Control guidance prior to Screening or must be negative for SARS-CoV-2 by polymerase chain reaction (PCR) within 72 hours of the Day 1 visit.
5. Body Mass Index (BMI) ≤34.9 kg/m2 and weight ≥50 kg.

Exclusion Criteria for SCD Participants

1. Evidence of ongoing uncontrolled clinically significant co-morbidity (e.g. intercurrent events that result in signs symptoms that have an adverse impact on the respective individual's usual function) hematological (non-SCD), renal, endocrine, pulmonary, gastrointestinal, cardiovascular (including stroke within 2 years prior to screening), hepatic, psychiatric or neurological.
2. Evidence or history of cardiac disease includes myocardial infarction, clinically significant cardiac arrhythmia (eg, atrial fibrillation, paroxysmal atrial fibrillation, atrial flutter, supraventricular tachycardia, and ventricular tachycardia), left ventricular failure, unstable angina, and coronary artery bypass grafting.
3. History of cancer (other than cutaneous basal cell or carcinoma in-situ) in the previous 5 years.
4. Active infection with Hepatitis B or C or HIV. Individuals seropositive for infection with Hepatitis C must be negative for viral RNA by PCR on at least 2 determinations.
5. History of active or latent tuberculosis (TB) regardless of treatment or positive QuantiFeron TB test.
6. Major surgery <3 months prior to baseline or planned significant medical procedures during the study.
7. Participants with any of the following acute or chronic infections or infection history:

   * Any infection requiring systemic treatment within 2 weeks prior to the screening visit.
   * Any infection requiring hospitalization, parenteral antimicrobial therapy within 30 days of the first dose of investigational product.
   * Any infection judged to be an opportunistic infection, within the past 6 months of the first dose of the investigational product.
   * Known active or history of frequent viral, fungal or other infections as determined by the Investigator.
   * Participants with a fever within the last 7 days prior to dosing.
8. Evidence or history of clinically significant orthostatic blood pressure changes.
9. Other acute or chronic medical or psychiatric condition that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
10. Participants with a history of allergic or anaphylactic reaction to therapeutic or diagnostic protein.
11. Administration of voxelotor within 4 weeks prior to screening or planned use during the study.
12. Administration of crizanlizumab within 12 weeks prior to screening or planned use during the study.
13. Planned transfusion during the study.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Frequency, severity and causal relationship of treatment emergent adverse events (TEAEs) and withdrawals due to TEAEs | Day 1 up to Day 85 (SAD) or Day 113 (MD)
  Frequency, severity and causal relationship of treatment emergent adverse events (TEAEs) and withdrawals due to TEAEs
Percentage of subjects with laboratory abnormalities | Day 1 up to Day 85 (SAD) or Day 113 (MD)
  Percentage of subjects with laboratory abnormalities
Number of subjects with change from baseline in vital signs | Day 1 up to Day 85 (SAD) or Day 85 (MD)
  blood pressure, pulse rate, temperature, respiration rate
Number of subjects with change from baseline in electrocardiogram (ECG) parameters | Day 1 up to Day 85 (SAD) or Day 85 (MD)
  Number of subjects with change from baseline in electrocardiogram (ECG) parameters
Percentage of subjects with injection site reactions | Day 1 up to Day 11 post (SAD) Day 1 up to Day 85 (MD)
  Percentage of subjects with injection site reactions
Percentage of subjects with infusion site reactions | Day 1 up to Day 11 post each dose (SD)
  Percentage of subjects with infusion site reactions

SECONDARY OUTCOMES:
SAD: Single Dose PK /Cmax | Day 1 up to Day 85
  Maximum serum concentration
SAD: Single Dose PK / DN Cmax | Day 1 up to Day 85
  Dose normalized Cmax
SAD: Single Dose PK / Tmax | Day 1 up to Day 85
  Time for Cmax
SAD: Single Dose PK / AUClast | Day 1 up to Day 85
  Area under the serum concentration time profile from time zero to the time of the last quantifiable concentration.
SAD: Single Dose PK / DN AUClast | Day 1 up to Day 85
  Dose normalized AUClast
SAD: Single Dose PK / AUCinf | Day 1 up to Day 85
  Area under the serum concentration time profile from time zero to infinity.
SAD: Single Dose PK / DN AUCinf | Day 1 up to Day 85
  Dose normalized AUCinf.
SAD: Single Dose PK / t½ | Day 1 up to Day 85
  Terminal half life
SAD: Single Dose PK / CL (IV only) | Day 1 up to Day 85
  Clearance
SAD: Single Dose PK / CL/F (SC only) | Day 1 up to Day 85
  Apparent clearance
SAD: Single Dose PK / Vss (IV only) | Day 1 up to Day 85
  Volume of distribution at steady state
SAD: Single Dose PK / Vz/F (SC only) | Day 1 up to Day 85
  Apparent volume of distribution at steady state
SAD: Single Dose PK / F (SC only) | Day 1 up to Day 85
  Apparent bioavailability
MD: AUCtau | Day 1 up to Day 22
  Area under the curve over the dosing interval tau (1 week) after the first and last doses
SAD:ADA and/or NAb | Day 1 up to Day 85
  Frequency of anti-drug antibody (ADA) and/or neutralizing antibody (NAb) productions
MD:ADA and/or NAb | Day 1 up to Day 113
  Frequency of anti-drug antibody (ADA) and/or neutralizing antibody (NAb) productions
Patient-reported VOC event rate and VOC day rate | Day 1 to 85
  Efficacy in SCD participants based on an electronic patient reported outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- United States (14):
  - New Haven Clinical Research Unit, New Haven, Connecticut
  - Howard University College of Medicine, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Lee Health - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Foundation for Sickle Cell Disease Research, Hollywood, Florida
  - Children's Healthcare of Atlanta - Egleston Hospital-Aflac Cancer and Blood Disorders Center, Atlanta, Georgia
  - University of Illinois at Chicago Clinical Research Center, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Prism Research LLC dba Nucleus Network, Saint Paul, Minnesota
  - Columbia University Medical Center - Herbert Irving Pavilion, New York, New York
  - CUIMC Research Pharmacy, New York, New York
  - CUMC Research Pharmacy, New York, New York
  - UT Physicians Comprehensive Sickle Cell Center Houston, Houston, Texas
  - Memorial Hermann clinical research unit, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4071001